CLINICAL TRIAL: NCT01276925
Title: The Effect of Ultrasound Guided Blockade of the Femoral Nerve, the Anterior Division of the Obturator Nerve, and the Lateral Femoral Cutaneous Nerve on Postoperative Pain, Morphine Consumption, and Mobilization After Total Hip Arthroplasty.
Brief Title: Total Hip Arthroplasty: Multiple Blocks by UltraSound
Acronym: THAMBUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Kenneth Jensen, MD, BBA, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBH-Z-THAMBUS
Record Dates: First submitted 2011-01-13; First posted 2011-01-14 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Pain, Postoperative
Keywords: Hip arthroplasty; Peripheral nervous blockade; Postoperative; Pain; Ropivacaine
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Ropivacaine; Ultrasonography; Sodium Chloride; Arthroplasty, Replacement, Hip; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- B3: Blockade of three nerves (Active Comparator): Peripheral nerve blockade of the femoral nerve, the anterior division of the obturator nerve, and the lateral femoral cutaneous nerve with ropivacaine.
  Interventions: Drug: Ropivacaine; Device: Ultrasound; Procedure: Peripheral nerve blockade; Procedure: Total hip arthroplasty; Drug: Bupivacaine
- B2: Blockade of 2 nerves (Active Comparator): Peripheral nerve blockade of the anterior division of the obturator nerve and the lateral femoral cutaneous nerve with ropivacaine.
  Sham blockade of the femoral nerve with saline.
  Interventions: Drug: Ropivacaine; Device: Ultrasound; Procedure: Peripheral nerve blockade; Drug: Saline; Procedure: Total hip arthroplasty; Drug: Bupivacaine
- K: Control group (Sham Comparator): Sham blockade of the femoral nerve, the anterior division of the obturator nerve, and the lateral femoral cutaneous nerve with saline.
  Interventions: Device: Ultrasound; Procedure: Peripheral nerve blockade; Drug: Saline; Procedure: Total hip arthroplasty; Drug: Bupivacaine

INTERVENTIONS:
Drug: Ropivacaine — 7,5 mg/ml. 10 ml for the femoral nerve, 10 ml for the anterior division of the obturator nerve, 5 ml for the lateral femoral cutaneous nerve.
  Other Names: Naropin
  Arms: B3: Blockade of three nerves
Drug: Ropivacaine — 7,5 mg/ml. 10 ml for the anterior division of the obturator nerve, 5 ml for the lateral femoral cutaneous nerve.
  Other Names: Naropin
  Arms: B2: Blockade of 2 nerves
Device: Ultrasound — All nerve blockades will be performed with ultrasound guidance.
Procedure: Peripheral nerve blockade — All patients will receive injections around the three nerves before surgery.
Drug: Saline — Isotonic. 10 ml for the femoral nerve.
  Arms: B2: Blockade of 2 nerves; K: Control group
Procedure: Total hip arthroplasty — All patients undergoes total hip arthroplasty.
Drug: Bupivacaine — 5 mg/ml. 3 ml for spinal anaesthesia.
  Other Names: Marcain spinal

SUMMARY:
Patients undergoing total hip arthroplasty may experience severe postoperative pain. This is normally treated with opioids, which can cause side effects such as nausea, vomiting, obstipation and sedation. The hypothesis is that patients receiving peripheral nerve blockade of three nerves leading pain stimuli from the hip will experience less pain, will consume less opioid and therefore have less side effects, and will be mobilized more quickly than patients not receiving the peripheral nerve blockade.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) may cause significant postoperative pain. The patients are often elderly, and frequently have other diseases or ailments. Postoperative pain treatment must focus on effective pain relief, keeping adverse effects to a minimum, enhancing physical rehabilitation and reducing postoperative morbidity.

Postoperative pain after hip surgery can be treated in different ways; i.e. paracetamol, NSAIDs, opioids, peripheral nerve blocks and epidural catheter. The choice seems to be influenced by local experience, education and personal preferences. Frequently, a multimodal approach is used with a combination of weak analgetics, opioids and maybe regional anaesthetic techniques.

The sensory innervation of the hip is through branches from the lumbar and sacral plexuses. The femoral nerve (FN), the obturator nerve (anterior branch) (ONA) and the lateral femoral cutaneous nerve (LCFN) all stem from the lumbar plexus. The FN and ONA directly supply the hip joint. LCFN innervates the skin on the lateral part of the thigh, where the incision for THA is often made.

The psoas compartment block provides good pain relief after THA, but the block can be associated with more frequent complications than other regional blockades for the lower extremity. Furthermore, the technique is difficult, and requires sub-specialized anaesthetists. In addition, it is often necessary to use electrical nerve stimulation together with ultrasound guidance to achieve a sufficient block.

Blockade of the FN is standard for hip fractures in our hospital, but not standard for THA. Because of the analgetic effect in hip fractures, the PROSPECT group recommends blockade of FN for THA as well, though specific evidence is scarce on the subject.

Blockade of the obturator nerve has been shown to provide pain relief for the hip joint, although the findings are not consistent, probably because of the varying innervation of the hip. The nerve is difficult to locate blindly, and location by nerve stimulator can be uncomfortable for the patient. Furthermore, the anatomic variations of the nerve and its branches is quite substantial.

Previously, nerves were located by surface anatomic landmarks or by nerve stimulation. In the past 6-7 years, the use of ultrasound guidance has become an increasingly effective aid for applying peripheral nerve blockades with continuingly improving technology.

Ultrasound-guided blockade of the three nerves (FN, ONA and LFCN) for postoperative pain treatment for THA is to our knowledge not previously described in the literature. From our knowledge of the anatomic course of the nerves, the investigators assume that the blockades can provide effective pain relief in this clinical context.

Our aim in this trial is to study the effect of ultrasound-guided periferal nerve blockade of the femoral nerve, the obturator nerve (anterior branch), and the lateral femoral cutaneous nerve on postoperative pain, opioid consumption and mobilization after THA.

The investigators want to describe the effect of blockade of the three nerves on pain, compared to placebo (injections with a well-known local analgesic drug compared to injections with isotonic saline).

Because it is desirable to have the patient mobilized as quickly as possible after operation, it seems optimal to cause as little motor blockade as possible. The investigators therefore also want to investigate whether pain relief with blockade of ONA and LCFN without blockade of FN is better than or equal to placebo.

The investigators want to study the possible differences in adverse effects, including motor blockade, between the groups with active nerve blockades, with and without blockade of FN.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years of age
* Patients scheduled for primary, unilateral hip arthroplasty with spinal anaesthesia
* Patients who have given their written and informed consent to participation after having understood the content and limitations of the protocol fully
* ASA 1-3

Exclusion Criteria:

* Patients who are not able to co-operate
* Patients who do not speak or understand Danish
* Daily use of opioids corresponding to 40 mg of morphine daily
* Allergy towards the drugs used in the study
* Drug abuse (investigators judgement)
* Alcohol consumption larger than advised by the Danish National Board of Health
* Spinal anaesthesia is contraindicated or the patient wants a general anaesthesia
* Patients in whom the blockade procedure or the spinal anaesthesia procedure cannot be completed because of technical difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2011-08; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Pain | At intervals during the first 48 hours after surgery
  Verbal Rating Scale score (0-10) at rest.

SECONDARY OUTCOMES:
Pain | At intervals during the first 48 hours after surgery
  Assessed by:
  * Verbal Rating Scale score (0-10) with passive flexion of the hip.
  * Verbal Rating Scale score (0-10) with active flexion of the hip.
Opioid consumption | In intervals during the first 48 hours after surgery
Bowel movement | Within the first 48 hours after surgery
  Assessed by:
  * Time for first stool
  * Number of stools at intervals during the first 48 hours after surgery
Sedation | At intervals during the first 48 hours after surgery
  Assessed by the Pasero Opioid-induced Sedation Scale (POSS).
Nausea | At intervals during the first 48 hours after surgery
  Assesed by
  * a verbal scale (none, light, moderate, marked)
  * the consumption of antiemetics
Vomiting | In intervals during the first 48 hours after surgery
  Number of vomitings, estimated to have exceeded a volume of 10 ml.
Mental and physical condition | Before and at intervals during the first 48 hours after surgery
  Assessed by:
  * Big Five Inventory, subscales extrovert and neuroticism
  * Modified Barthel Index/100
  * SF-8 index
Mobilization | The first 48 hours after surgery
  The time at which the patient walks for the first time after surgery.
Length of stay | One week
  * The time from end of surgery to discharge from the postoperative care unit
  * The time from end of surgery to discharge from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte M Krogh, MD, Principal Investigator — Bispebjerg Hospital; Kenneth Jensen, MD, Study Director — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark